CLINICAL TRIAL: NCT02758340
Title: Comparison of Maternal Outcome Between Patients Undergoing Induction of Labor With Oral Misoprostol Alone and Oral Misoprostol and Foley's Catheter Both at a Tertiary Care Hospital
Brief Title: Failure of Vaginal Delivery After Induction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karachi Medical and Dental College (Other)
Responsible Party: Principal Investigator, samia husain, postgraduate trainee, Karachi Medical and Dental College
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: KarachiDMC
Record Dates: First submitted 2016-04-27; First posted 2016-05-02 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Labor Pain
Keywords: induction of labor; misoprostol; foley's balloon catheter
MeSH Terms: conditions — Labor Pain | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- M=misoprostol (Experimental): Patients who would receive Only oral misoprostol{(50 micrograms) tab cytotec ¼ tablets (Searle)}. All patients in this group will be given oral misoprostol 50 μg per dose. The dose will be repeated at 4 hours interval up to a maximum of 4 doses till labor is induced (3 contractions per 10 minutes). If labor is not established within 4 hours of the administration of the fourth dose, induction will be considered to be failed
  Interventions: Drug: Misoprostol
- M+F=MISOPROSTOL+FOLEY'S BALLOON CATHETER (Experimental): All patients in this group will be explained the technique of foley's catheter ballooning and informed consent will be taken. The cervix will be visualized with the help of Cusco's speculum. The balloon will be inflated with about 30 cc of sterile water. The catheter will be pulled down to bring the balloon into the cervical canal and will be tapped around the thigh. Patients will also be given oral misoprostol 50 μg per dose. The dose will be repeated at 4 hours interval up to a maximum of 4 doses till labor is induced (3 contractions per 10 minutes).
  Interventions: Drug: Misoprostol; Device: foley's balloon catheter

INTERVENTIONS:
Drug: Misoprostol — Women would be given misoprostol tablet by mouth
  Other Names: cytotec
Device: foley's balloon catheter — foley's balloon catheter would be inserted through vagina into cervix.
  Other Names: foley's catheter
  Arms: M+F=MISOPROSTOL+FOLEY'S BALLOON CATHETER

SUMMARY:
The study will compare the number of women who deliver vaginally after artificial initiation of labor pains(i.e. induction of labor) by two methods. Half of the women would receive tablet misoprostol vaginally and the other half would receive tablet misoprostol and foley's balloon catheter both.

DETAILED DESCRIPTION:
Artificial initiation of labor pains has become a common occurrence. A variety of methods are employed to initiate labor pains. Labor pains are more successful in culminating into vaginal delivery if the neck of womb that is the cervix is soft (ripe). This is usually achieved by ripening agents. They include drugs and devices that help soften the cervix. Misoprostol and foley's balloon catheter both are used to soften the cervix so that vaginal delivery is possible. Both work on different aspects of the softening of cervix.

Misoprostol acts on shortening the cervix and making it more pliable Foley's balloon helps to open up the cervix that is it aids in dilating the cervical canal.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 37 weeks assessed by Last Menstrual Period and dating scan.
* Women with singleton pregnancy assessed by ultrasound.
* Fetus in vertex presentation assessed by ultrasound.
* Age 20-40 years.
* Bishop score <4.

Exclusion Criteria:

* Non-consenting.
* Gestational age < 37 weeks.
* Patients with history of placenta previa.
* Patients with history of placental abruption.
* Ruptured membranes.
* Patients with history of vaginal infection.
* Patients with history of congenital anomalies in previous deliveries.
* Patients with history of stroke, renal impairment and chronic obstructive pulmonary disease, chronic liver disease and congestive cardiac failure

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 335 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
failure of vaginal delivery i.e.percentage of women in both groups who would fail to deliver vaginally after 24 hours of induction. | six months

CONTACTS AND LOCATIONS:
Overall Officials: samia husain, MBBS, Principal Investigator — Karachi Medical and Dental College
Locations (1):
- Abbasi shaheed hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264